CLINICAL TRIAL: NCT02774356
Title: Testing Native Language Neural Commitment at the Subcortical Level: Links Between Brainstem Frequency Following Responses and Behavioral Perception for Lexical Tones
Brief Title: Testing Native Language Neural Commitment at the Subcortical Level
Status: Completed | Type: Observational
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Other Study IDs: 1505M69162
Record Dates: First submitted 2015-06-09; First posted 2016-05-17 (Estimated); Last update posted 2017-01-18 (Estimated); Status verified 2017-01

CONDITIONS: Language Development
Keywords: Brainstem; Encoding; Pitch

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Native Chinese speakers
- Native English speakers without experience of a tonal language

SUMMARY:
This mentored student research project is funded by the Graduate Research Partnership Program with a projected timeline for data collection in the summer of 2015. Previous research has shown that language experience alters the way the human brain processes speech information. This phenomenon takes place very early in life and is referred to as Native Language Neural Commitment. For instance, as the Japanese language does not have the l-r speech sound contrast, Japanese infants start to show difficulty in hearing differences between the English l and r sounds at 12 months of age but not when they were at 6 months old. Learning the l-r distinction later in life proves to be very difficult for the Japanese school students and adults. Brain imaging studies have further revealed specific brain regions that are changed by language learning. But the evidence in support of the Native Language Neural Commitment theory is based on cortical-level measures. The proposed study extends the measurement to the subcortical level at the brainstem. The target language that the investigators are interested in studying is Mandarin Chinese, which is known for its use of lexical tones to express different words. For instance, the Chinese syllable "ma" means "mother" when it is spoken with a flat tone, and it means "hemp" when spoken with a rising tone. English, by contrast, does not employ lexical tones, and it is considered a non-tonal language. Does the Chinese learning experience fundamental change the way that pitch information is coded in the human brain? Does it happen at both cortical and subcortical levels? Previous research has shown evidence for a positive answer to both questions. But the direct evidence for brain-behavior correlations at the subcortical level is still missing.

The proposed cross-language study will test Chinese-speaking and English-speaking adults to investigate Native Language Neural Commitment at the subcortical level. The investigators are interested in differences in the two subject populations by examining the relationship between brainstem pitch tracking and behavioral pitch perception in linguistic and nonlinguistic stimuli.

The results of the proposed project will contribute to the understanding the role of the subcortical brainstem in Native Language Neural Commitment, which have significant implications for the development of auditory/speech training programs and assessment tools utilizing the brainstem frequency following measure to monitor progress in second language learning and test clinical populations.

ELIGIBILITY:
Inclusion Criteria:

1. Native Mandarin Chinese speakers
2. Native English speakers
3. Non-musicians.
4. English speakers must have no prior experience with a tonal language.
5. Normal hearing
6. Age range to 18-50.

Exclusion Criteria:

1. Speech-language-hearing disorders, neurophysiological/psychiatric conditions, including stroke or brain injuries, which would prevent the subject from sitting still and performing the experimental tasks.
2. Subjects with three or more than three years of musical practice/training will be excluded.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Normal healthy adult population.
Sampling Method: Non-Probability Sample
Enrollment: 36 (Actual)
Dates: Start 2015-07; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Pitch strength of Brainstem EEG (electroencephalography) responses | Outcome will be measured at one 1.5-hr session after the participant is recruited.
  EEG signals to pitch changes in speech and nonspeech sounds are analyzed to obtain the brainstem frequency following responses (FFRs). Autocorrelation method will be applied to the FFRs to quantify each participant's brainstem pitch strength. Higher average autocorrelation value indicates greater pitch strength. This EEG measure is to see whether tonal-language speakers and nontonal language speakers differ in brainstem encoding of pitch information.
Reaction time in millesecond for speech perception of syllables with varying pitch contour | Outcome will be measured at one 1.5-hr session after the participant is recruited.
  This behavioral measure in terms of syllable perception is to test whether syllabic perception is influenced by pitch information and whether tonal-language speakers' sensitivity towards pitch differences would affect the speech perception differently.
Correlation between the EEG and the Behavioral measures | Outcome will be measured at one 1.5-hr session after the participant is recruited.
Pitch tracking accuracy of Brainstem EEG (electroencephalography) responses | Outcome will be measured at one 1.5-hr session after the participant is recruited.
  Strength of stimulus-to-response correlation will assessed. Higher correlation coefficient between the fundamental frequency of the stimulus and that of the FFR response will indicate greater accuracy of the brainstem pitch tracking. This EEG measure is to see whether tonal-language speakers and nontonal language speakers differ in brainstem encoding of pitch information.
Duration estimate of syllables with varying pitch contour | Outcome will be measured at one 1.5-hr session after the participant is recruited.
  This behavioral measure in terms of syllable duration estimation is to test whether duration estimation is influenced by pitch information and whether tonal-language speakers' sensitivity towards pitch differences would affect the duration estimation differently.

CONTACTS AND LOCATIONS:
Locations (1):
- Zhang Lab at Department of Speech-Language-Hearing Sciences, Minneapolis, Minnesota, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Krishnan A, Xu Y, Gandour J, Cariani P. Encoding of pitch in the human brainstem is sensitive to language experience. Brain Res Cogn Brain Res. 2005 Sep;25(1):161-8. doi: 10.1016/j.cogbrainres.2005.05.004. PMID 15935624
- [Background] Zhang Y, Kuhl PK, Imada T, Kotani M, Tohkura Y. Effects of language experience: neural commitment to language-specific auditory patterns. Neuroimage. 2005 Jul 1;26(3):703-20. doi: 10.1016/j.neuroimage.2005.02.040. Epub 2005 Apr 13. PMID 15955480
- [Background] Bidelman GM, Gandour JT, Krishnan A. Musicians and tone-language speakers share enhanced brainstem encoding but not perceptual benefits for musical pitch. Brain Cogn. 2011 Oct;77(1):1-10. doi: 10.1016/j.bandc.2011.07.006. Epub 2011 Aug 10. PMID 21835531
- [Background] Marmel F, Linley D, Carlyon RP, Gockel HE, Hopkins K, Plack CJ. Subcortical neural synchrony and absolute thresholds predict frequency discrimination independently. J Assoc Res Otolaryngol. 2013 Oct;14(5):757-66. doi: 10.1007/s10162-013-0402-3. Epub 2013 Jun 13. PMID 23760984
- [Background] Xu Q, Gong Q. Frequency difference beyond behavioral limen reflected by frequency following response of human auditory Brainstem. Biomed Eng Online. 2014 Aug 9;13:114. doi: 10.1186/1475-925X-13-114. PMID 25108552